CLINICAL TRIAL: NCT06439797
Title: Inflammatory Markers as Predictors of the Efficacy of Electroconvulsive Therapy (ECT) in Major Depression Patients
Acronym: ECT MDD
Status: Completed | Type: Observational
Sponsor: The Chaim Sheba Medical Center (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Principal Investigator, Revital Amiaz, Head of Psychiatry Department B, The Chaim Sheba Medical Center, Tel Aviv University
Other Study IDs: 5040-18-SMC
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder; Healty Controls
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: ECT is an effective treatment indicated for patients with treatment resistant depression. Although most patients display some degree of recovery, 32-52% do not respond or remit at all. Considering the possible side effects and the considerably high cost of treatment, it is important to identify sub-populations that would benefit the most from ECT. In the current study we sought to identify predictive molecular markers in the blood of depressed patients who are responsive to ECT.

Methods: Patients, ages 18-70, with the diagnosis of treatment-resistant depression will be recruited. Participants will undergo psychiatric and psychological assessments, before (baseline) and 12 weeks after ECT initiation. Assessments will include the Montgomery-Asberg Depression Rating Scale (MADRAS), Clinical Global Improvement and Severity Scales (CGI-S, CGI-I), Inventory of Depressive Symptomatology (IDS), and the State-Trait Anxiety Inventory (STAI). Blood samples for serum and isolation of peripheral blood mononuclear cells (PBMCs)will be collected at baseline and the 12-week end-of-treatment time points for molecular analysis.

DETAILED DESCRIPTION:
Despite impressive progress in our understanding of the molecular, cellular and circuit-level correlates of major depression, the biological mechanisms that causally underlie this disorder remain unclear, hindering the development of effective novel therapeutic procedures. One possible reason for this situation is that almost all research in this area focuses on the involvement of abnormalities in neuronal functioning, whereas the involvement of non-neuronal brain cells, particularly microglia, has not been thoroughly investigated. Recent studies indicate that impairments of the normal structure and function of microglia, caused by either intense inflammatory activation or by decline and senescence of these cells, can lead to depression and associated impairments in neuroplasticity and neurogenesis. Accordingly, we argued that at least some forms of depression can be considered as microgliopathies, in which either microglial activation or microglial decline and suppression constitute the direct etiology of the depressive syndrome. This implies that depression cannot be treated uniformly but should rather be treated by a personalized medical approach based on the microglial status of the individual depressed patient (Yirmiya et al., TiNS, 2015). In the current proposal we aim to lay foundations for a thorough examination of the personalized medical approach to depression, by examining the benefits of personalized utilization of anti-depressive procedures based on screening for inflammatory/ microglial markers, and by developing state-of-the-art tools for microglia manipulations that will allow to directly examine the causal role of these cells in various animal models of depression.

We specifically aim to develop a personalized approach to the utilization of electroconvulsive therapy (ECT), because our preliminary findings in a mouse model of depression associated with impaired microglia functioning conclusively show that ECT-induced microglia activation is causally related to the anti-depressive effects of this treatment. We propose to utilize a translational approach, assessing the inflammatory/microglia-related molecular factors (measured before treatment) that predict and contribute to the efficacy of ECT in major depression patients. Specifically, we expect that ECT will be more beneficial in patients with low expression of inflammatory/microglia-related genes, and thus based on the findings of this experiment we shall be able to devise a molecular screening for the suitability of ECT (and possibly other anti-depressant procedures) for the individual depressed patient. Furthermore, we aim to establish the transcriptomic effects of ECT, with a particular emphasis on inflammatory-related pathways. We expect differential transcriptomic effects of ECT in patients with high vs. low baseline inflammatory status. The results should significantly contribute to our knowledge regarding the molecular mechanisms that underlie the therapeutic effects of ECT in specific sub-groups of depressed patients.

In parallel studies we aim to develop molecular tools for selective and region-specific microglia activation or inhibition and to use these tools for: 1) examining the effects of these manipulations in animal models of depression that involve either hyper-or hypo-activity of microglia. 2) defining the causal role of microglia in mediating the anti-depressive effects of ECT in a depression model associated with low microglia status. These studies should complement the clinical part in humans, by providing definitive evidence for the inverted U-shape pattern of relations between inflammatory status and depression, which constitutes the basis for the personalized medical approach to this disease.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to provide informed consent. Able to adhere to the treatment schedule. Are treated for the current depressive episode, at least four weeks, with at least one antidepressant in accepted dose, without improvement, according to their medical chart and ATHF (antidepressant treatment history form) instruction guidelines.

Exclusion Criteria:

* Diagnosis of an autoimmune disease. History of disturbances with bone marrow functioning. History of Oncologic Diseases. History of drug abuse or alcoholism in the last 6 months. Suffering from another diagnosis on axis 1, including schizophrenia, and geriatric depression.

Patients with any current unstable medical illness. Any condition involving fluid retention, pulmonary infiltrates, congestive heart failure, respiratory symptoms or disease, cardiac symptoms or disease, and renal or hepatic dysfunction Patients taking lithium or corticosteroids. Pregnancy or not using a reliable method of birth control. Neurodegenerative diseases (i.e: Alzheimer's disease, Parkinson's disease). Participation in a current interventional clinical study or interventional clinical study within 30 days before this study.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major Depressive Disorder with treatment-resistant disorder referred to the ECT clinic
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-11-29 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Inflammatory Markers as Predictors of the efficacy of Electroconvulsive Therapy (ECT) in Major Depression Patients. | Before ECT treatment and after 12 treatments, After 3 weeks
  Patients, ages 18-70, with the diagnosis of treatment-resistant depression will recruited. Participants will undergo psychiatric and psychological assessments, before (baseline) and 12 weeks after ECT initiation. Assessments included the Montgomery-Asberg Depression Rating Scale (MADRAS), Clinical Global Improvement and Severity Scales (CGI-S, CGI-I), Inventory of Depressive Symptomatology (IDS), and the State-Trait Anxiety Inventory (STAI). Blood samples for serum and isolation of peripheral blood mononuclear cells (PBMCs) will be collected at baseline and the 12 weeks end-of-treatment time points for molecular analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Revital Amiaz, Ramat Gan, RI, Israel